CLINICAL TRIAL: NCT06404489
Title: Evaluation of a Multimodal Program of Prehabilitation in Oncological Patients Undergoing Major Gastrointestinal Surgery Within an ERAS Pathway.
Brief Title: Prehabilitation in Oncological Patients Undergoing Major Gastrointestinal Surgery (PROGRESS)
Acronym: PROGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROGRESS - CET 191-2023
Record Dates: First submitted 2024-04-24; First posted 2024-05-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Oncological Patients; Major Surgery
Keywords: Prehabilitation; Multimodal prehabilitation program; Standard care treatment; Major gastrointestinal surgery; Hospital stay; Functional walking; Nutrition; Diet; Exercise; Relaxation; Oncology; Functional recovery; Anesthesiology
MeSH Terms: conditions — Motor Activity; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Prehabilitation arm group will receive preoperative intervention which includes exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline.
  Interventions: Behavioral: Multimodal prehabilitation Program
- Control group (No Intervention): Standard care treatment. Application of ERAS pathways (Enhanced Recovery After Surgery)

INTERVENTIONS:
Behavioral: Multimodal prehabilitation Program — A tailored intervention will be prescribed if specific physical, nutritional or psychological impairments will be identified during the assessment phase. Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, and/or nutrition optimization, and/or distress-coping techniques. Different combinations of three domains will be utilized to maximize their synergistic anabolic effect.
  The duration of program will be set at 4 weeks. All activities will be performed in dedicated suites at each site, under supervision of qualified health professionals.
  Arms: Prehabilitation

SUMMARY:
The importance of postoperative rehabilitation on physical performance and recovery is well-recognized. However, the preoperative period constitutes a unique opportunity to address comorbidities and modifiable risk factors, improve functional capacity and address deficiencies in physiologic reserve, which might otherwise preclude surgery or significantly impede recovery.

Therefore, the aim of this study is to evaluate the efficacy of a multimodal program of prehabilitation in patients undergoing major oncological gastrointestinal surgery. The hypothesis is that severe post-operative complications within 30 days will be reduced in the treatment group compared to the control group.

DETAILED DESCRIPTION:
This is a 2-arm randomized multicentric controlled trial to test the efficacy of a personalized, multidisciplinary, preoperative conditioning program to reduce severe complications and facilitate recovery in patients undergoing major oncological gastrointestinal surgery.

400 patients will be randomized (ratio 1:1) and allocated either to the intervention group (Prehabilitation), or to the control group (which will be treated according to usual standard of care within Enhanced Recovery After Surgery (ERAS) pathways).

Multimodal prehabilitation is a preoperative intervention which includes exercise training, nutritional therapy and anxiety reducing techniques, aimed at preventing or attenuating surgery-driven functional decline.

The primary objective is to evaluate the effect of a multimodal program of prehabilitation on postoperative severe complications.

Secondary outcomes include time to functional recovery, length of hospital stay, complication severity, proportion of patients returning to preoperative functional walking capacity and self-reported activity status and generic health related quality of life at 30 days after surgery.

Included patients will be randomized and allocated either to the intervention group, which will receive 4 weeks of prehabilitation, or to the control group, which will receive no prehabilitation. All patients will be reassessed the day before surgery, 30 days and 3 months after surgery.

Patients enrolled in treatment group will not receive any additional medication but only a multimodal program to optimize their preoperative functional capacity.

Within 30 days prior to scheduled surgery, participants of both groups will undergo a specialized multidisciplinary assessment with a physician, a certified physiotherapist, registered dietitian and psychology trained personnel. All tests will be performed following international guidelines and standardized verbal instructions. A tailored intervention will be prescribed if specific physical, nutritional or psychological impairments will be identified during the assessment phase. Based on the data obtained during the multimodal assessment, different domains and levels of care will be prescribed, focusing on exercise training, and/or nutrition optimization, and/or distress-coping techniques. Different combinations of three domains will be utilized to maximize their synergistic anabolic effect.

Statistical analysis will be performed according to study sites, type of surgery (esophageal, gastric, colonic, rectal) and neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age > 18 years) scheduled for elective gastrointestinal surgery for cancer.
* Signed informed consent

Exclusion Criteria:

Co-morbid medical, physical, and mental conditions interfering with the ability to complete study procedures, such as:

* acute or unstable cardio-respiratory conditions (e.g., unstable angina or symptomatic severe aortic stenosis)
* severe/end-stage organ diseases (e.g., cardiac failure NYHA functional classes III-IV, COPD FEV1 <50% pred, end-stage kidney or liver disease);
* American Society of Anesthesiologists (ASA) physical status classes 4-5.
* disabling orthopedic and neuromuscular disease.
* psychosis, dementia;
* symptomatic anemia.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | Evaluation of severe post-operative complications within 30 days
  Reduction of incidence of postoperative complications.

SECONDARY OUTCOMES:
Lenght of hospital stay | 30 days after surgery
  Reduction of lenght of hospital stay in treatment group
Proportion of patients returning to preoperative functional walking capacity | 30 days after surgery, 90 days follow up after surgery
  Improving return to basal functional preoperative capacity

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria, Cagliari, Sardinia
  - IRCCS San Raffaele Scientific Institute, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Bautmans I, Njemini R, De Backer J, De Waele E, Mets T. Surgery-induced inflammation in relation to age, muscle endurance, and self-perceived fatigue. J Gerontol A Biol Sci Med Sci. 2010 Mar;65(3):266-73. doi: 10.1093/gerona/glp145. Epub 2009 Oct 6. PMID 19808837
- [Background] Carli F. Physiologic considerations of Enhanced Recovery After Surgery (ERAS) programs: implications of the stress response. Can J Anaesth. 2015 Feb;62(2):110-9. doi: 10.1007/s12630-014-0264-0. Epub 2014 Dec 12. PMID 25501695
- [Background] Lemanne D, Cassileth B, Gubili J. The role of physical activity in cancer prevention, treatment, recovery, and survivorship. Oncology (Williston Park). 2013 Jun;27(6):580-5. PMID 23909073
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Shen Y, Hao Q, Zhou J, Dong B. The impact of frailty and sarcopenia on postoperative outcomes in older patients undergoing gastrectomy surgery: a systematic review and meta-analysis. BMC Geriatr. 2017 Aug 21;17(1):188. doi: 10.1186/s12877-017-0569-2. PMID 28826406
- [Background] Jack S, West MA, Raw D, Marwood S, Ambler G, Cope TM, Shrotri M, Sturgess RP, Calverley PM, Ottensmeier CH, Grocott MP. The effect of neoadjuvant chemotherapy on physical fitness and survival in patients undergoing oesophagogastric cancer surgery. Eur J Surg Oncol. 2014 Oct;40(10):1313-20. doi: 10.1016/j.ejso.2014.03.010. Epub 2014 Mar 27. PMID 24731268
- [Background] Carlsson E, Berndtsson I, Hallen AM, Lindholm E, Persson E. Concerns and quality of life before surgery and during the recovery period in patients with rectal cancer and an ostomy. J Wound Ostomy Continence Nurs. 2010 Nov-Dec;37(6):654-61. doi: 10.1097/WON.0b013e3181f90f0c. PMID 21052026
- [Background] Silver JK, Baima J. Cancer prehabilitation: an opportunity to decrease treatment-related morbidity, increase cancer treatment options, and improve physical and psychological health outcomes. Am J Phys Med Rehabil. 2013 Aug;92(8):715-27. doi: 10.1097/PHM.0b013e31829b4afe. PMID 23756434
- [Background] Wijeysundera DN, Pearse RM, Shulman MA, Abbott TEF, Torres E, Ambosta A, Croal BL, Granton JT, Thorpe KE, Grocott MPW, Farrington C, Myles PS, Cuthbertson BH; METS study investigators. Assessment of functional capacity before major non-cardiac surgery: an international, prospective cohort study. Lancet. 2018 Jun 30;391(10140):2631-2640. doi: 10.1016/S0140-6736(18)31131-0. PMID 30070222
- [Background] Pecorelli N, Fiore JF Jr, Gillis C, Awasthi R, Mappin-Kasirer B, Niculiseanu P, Fried GM, Carli F, Feldman LS. The six-minute walk test as a measure of postoperative recovery after colorectal resection: further examination of its measurement properties. Surg Endosc. 2016 Jun;30(6):2199-206. doi: 10.1007/s00464-015-4478-1. Epub 2015 Aug 27. PMID 26310528
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Boshier PR, Heneghan R, Markar SR, Baracos VE, Low DE. Assessment of body composition and sarcopenia in patients with esophageal cancer: a systematic review and meta-analysis. Dis Esophagus. 2018 Aug 1;31(8). doi: 10.1093/dote/doy047. PMID 29846548
- [Background] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Background] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805
- [Background] Zopfs D, Theurich S, Grosse Hokamp N, Knuever J, Gerecht L, Borggrefe J, Schlaak M, Pinto Dos Santos D. Single-slice CT measurements allow for accurate assessment of sarcopenia and body composition. Eur Radiol. 2020 Mar;30(3):1701-1708. doi: 10.1007/s00330-019-06526-9. Epub 2019 Nov 27. PMID 31776743
- [Background] Carli F, Gillis C, Scheede-Bergdahl C. Promoting a culture of prehabilitation for the surgical cancer patient. Acta Oncol. 2017 Feb;56(2):128-133. doi: 10.1080/0284186X.2016.1266081. Epub 2017 Jan 9. PMID 28067101
- [Background] Colado JC, Pedrosa FM, Juesas A, Gargallo P, Carrasco JJ, Flandez J, Chupel MU, Teixeira AM, Naclerio F. Concurrent validation of the OMNI-Resistance Exercise Scale of perceived exertion with elastic bands in the elderly. Exp Gerontol. 2018 Mar;103:11-16. doi: 10.1016/j.exger.2017.12.009. Epub 2017 Dec 17. PMID 29262307
- [Background] Babic B, Tagkalos E, Gockel I, Corvinus F, Hadzijusufovic E, Hoppe-Lotichius M, Lang H, van der Sluis PC, Grimminger PP. C-reactive Protein Levels After Esophagectomy Are Associated With Increased Surgical Trauma and Complications. Ann Thorac Surg. 2020 May;109(5):1574-1583. doi: 10.1016/j.athoracsur.2019.12.016. Epub 2020 Jan 24. PMID 31987821
- [Background] Schulz SVW, Schumann U, Otto S, Kirsten J, Treff G, Janni W, Huober J, Leinert E, Steinacker JM, Bizjak DA. Two-year follow-up after a six-week high-intensity training intervention study with breast cancer patients: physiological, psychological and immunological differences. Disabil Rehabil. 2022 Aug;44(17):4813-4820. doi: 10.1080/09638288.2021.1921861. Epub 2021 May 11. PMID 33974472
- [Derived] Oliva FM, Turi S, Veneziano M, D'Amico F, Passuello N, Notarianni L, Fiorindi C, De Piccoli N, Ripamonti L, Fossati L, Gualtierotti M, Ghezzi M, Vecchiato M, Pontillo D, Priolo S, Marchetti C, Sandona D, Cicero P, Nicastro V, Fumagalli A, Sarzo G, Kozhan P, Pecorelli N, Pieri M, Puccetti F, Foti S, Tettamanti A, Palumbo D, Basile G, Marmiere M, Fresilli S, Labanca R, Pruna A, Pasin L, Putzu A, Garcia CSR, Donadello K, Sardo S, Bove T, Nespoli L, Baldini G, Finco G, Vignali A, Beretta L; PROGRESS Study Group. Prehabilitation in oncological patients undergoing major gastrointestinal surgery: rationale and design of the PROGRESS trial. Contemp Clin Trials. 2026 Jan 30:108249. doi: 10.1016/j.cct.2026.108249. Online ahead of print. PMID 41621468